CLINICAL TRIAL: NCT02473640
Title: A Phase 1b/2a, Multi-Center, Open-Label, 2-Period, Fixed-Sequence Study Evaluating the Effect of Esomeprazole on SYN-004 Degradation of Ceftriaxone In Healthy Adult Subjects With a Functioning Ileostomy
Brief Title: A Study Evaluating the Effect of Esomeprazole on SYN-004 Degradation of Ceftriaxone In Adults With an Ileostomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theriva Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-1-004-004
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers With Ileostomy
MeSH Terms: interventions — SYN-004; Esomeprazole; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 150 mg SYN-004 (Experimental): There will be 2 in-house treatment periods: in Treatment Period 1, subjects will receive 2 oral doses of 150 mg SYN-004 (two 75 mg capsules) and 1g ceftriaxone, and in Treatment Period 2, subjects will receive 2 oral doses of 150mg SYN-004 (two 75 mg capsules) and 1g ceftriaxone in the presence of steady-state esomeprazole; Treatment Periods 1 and 2 will be separated by a 5- to 7-day run-in phase, during which subjects will self-administer 40 mg of esomeprazole once daily (QD) in the morning, at home.
  Interventions: Drug: SYN-004; Drug: Esomeprazole; Drug: Ceftriaxone

INTERVENTIONS:
Drug: SYN-004
Drug: Esomeprazole
Drug: Ceftriaxone

SUMMARY:
A Phase 1b/2a, Multi-Center, Open-Label, 2-Period, Fixed-Sequence Study Evaluating the Effect of Esomeprazole on SYN-004 Degradation of Ceftriaxone In Healthy Adult Subjects with a Functioning Ileostomy

DETAILED DESCRIPTION:
This is a Phase 1b/2a, randomized, multi-center, open-label study. Twenty otherwise healthy subjects with functioning ileostomies who are between the ages of 18 and 80 years, inclusive, will be enrolled. The entire duration of the study may be up to 63 days (from Screening to the end-of-study [EOS] visit).

ELIGIBILITY:
Inclusion Criteria:

* The subject has a functioning ileostomy that has been in place for ≥ 3 months.
* The subject is male or female between the ages of 18 and 80 years, inclusive.
* Other than a functioning ileostomy, the subject is free from clinically significant illnesses or disease.

Exclusion Criteria:

* Subjects who have active hepatic, small intestine, or biliary tract disease.
* Subjects who have active ulcerative colitis, Crohn's disease, other inflammatory bowel disease.
* Subjects with known malignancy requiring treatment < 6 months prior to study screening.
* Subjects who have, in the opinion of the investigator, significant concurrent medical illness.
* Subjects who are currently taking concomitant medications which may interfere with study evaluation.
* Subjects who have received an investigational drug within 30 days or within a time period consistent with a washout period of 5 half-lives, whichever is longer, of the first dose of ceftriaxone.
* Subjects with a known history of allergy to any cephalosporin, penicillin or any β-lactam antibiotic.
* Subjects who have known active malabsorption syndromes(s) that, in the judgment of the investigator, could compromise the objectives of the study.
* Subjects who have used any oral, intramuscular, or IV anti-microbial medication during the last 3 week

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Synthetic Biologics Investigative Site, Edmonton, Alberta
  - Synthetic Biologics Investigative Site, Montreal

REFERENCES:
- [Derived] Kokai-Kun JF, Roberts T, Coughlin O, Sicard E, Rufiange M, Fedorak R, Carter C, Adams MH, Longstreth J, Whalen H, Sliman J. The Oral beta-Lactamase SYN-004 (Ribaxamase) Degrades Ceftriaxone Excreted into the Intestine in Phase 2a Clinical Studies. Antimicrob Agents Chemother. 2017 Feb 23;61(3):e02197-16. doi: 10.1128/AAC.02197-16. Print 2017 Mar. PMID 28052855

RESULTS

PARTICIPANT FLOW:
Groups:
- 150 mg SYN-004: There will be 2 in-house treatment periods: in Treatment Period 1, subjects will receive 2 oral doses of 150 mg SYN-004 (two 75 mg capsules) and 1g ceftriaxone, and in Treatment Period 2, subjects will receive 2 oral doses of 150mg SYN-004 (two 75 mg capsules) and 1g ceftriaxone in the presence of esomeprazole; Treatment Periods 1 and 2 will be separated by a 5- to 7-day run-in phase, during which subjects will self-administer 40 mg of esomeprazole once daily (QD) in the morning, at home.
  SYN-004
  Esomeprazole
  Ceftriaxone
Period: Treatment Period 1
Arm/Group | 150 mg SYN-004
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1
Period: Run-in Phase
Arm/Group | 150 mg SYN-004
Started | 14
Completed | 14
Not Completed | 0
Period: Treatment Period 2
Arm/Group | 150 mg SYN-004
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 150 mg SYN-004: There will be 2 in-house treatment periods: in Treatment Period 1, subjects will receive 2 oral doses of 150 mg SYN-004 (two 75 mg capsules) and 1g ceftriaxone, and in Treatment Period 2, subjects will receive 2 oral doses of 150mg SYN-004 (two 75 mg capsules) and 1g ceftriaxone in the presence of steady-state esomeprazole; Treatment Periods 1 and 2 will be separated by a 5- to 7-day run-in phase, during which subjects will self-administer 40 mg of esomeprazole once daily (QD) in the morning, at home.
  SYN-004
  Esomeprazole
  Ceftriaxone
Arm/Group | 150 mg SYN-004
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Ceftriaxone Concentration in Intestinal Chyme Period 1
Description: Ceftriaxone concentration in the presence of SYN-004 and the absence of esomeprazole.
Time Frame: 0-8.5 hours
Population: Subjects with functioning illeostomies who received a single IV infusion of 1 g ceftriaxone.
Measure: Mean (Standard Error); unit: ug/mL
Groups:
- 150 mg SYN-004: There will be 2 in-house treatment periods: in Treatment Period 1, subjects will receive 2 oral doses of 150 mg SYN-004 (two 75 mg capsules) and 1g ceftriaxone, and in Treatment Period 2, subjects will receive 2 oral doses of 150mg SYN-004 (two 75 mg capsules) and 1g ceftriaxone in the presence of esomeprazole; Treatment Periods 1 and 2 will be separated by a 5- to 7-day run-in phase, during which subjects will self-administer 40 mg of esomeprazole once daily (QD) in the morning, at home.
Arm/Group | 150 mg SYN-004
Number analyzed (Participants) | 14
ug/mL
  Hour 0 | 0.00 (0.00)
  Hour 0.5 | 0.00 (0.00)
  Hour 1.5 | 5.60 (4.39)
  Hour 2.5 | 150.90 (68.43)
  Hour 3.5 | 231.40 (144.06)
  Hour 4.5 | 173.00 (98.58)
  Hour 5.5 | 29.00 (25.40)
  Hour 6.5 | 1.40 (0.82)
  Hour 7.5 | 0.10 (0.10)
  Hour 8.5 | 2.00 (1.70)

2. Primary Outcome: Ribaxamase Concentration in Intestinal Chyme Period 1
Description: Concentrations of ribaximase (SYN-004) in intestinal chyme
Time Frame: 0-8.5 hours
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | 150 mg SYN-004
Number analyzed (Participants) | 14
ng/mL
  Hour 0 | 0.00 (0.00)
  Hour 0.5 | 2 (2.1)
  Hour 1.5 | 11 (9.1)
  Hour 2.5 | 131 (116.8)
  Hour 3.5 | 6727 (3983.1)
  Hour 4.5 | 56795 (25155.4)
  Hour 5.5 | 73090 (29292.8)
  Hour 6.5 | 103171 (52510.2)
  Hour 7.5 | 153274 (87804.1)
  Hour 8.5 | 111946 (71722.7)

3. Primary Outcome: Ceftriaxone Concentration in Intestinal Chyme Period 2
Description: Ceftriaxone concentration in the presence of SYN-004 and the absence of esomeprazole.
Time Frame: 0-8.5 hours
Population: Subjects with functioning illeostomies who received a single IV infusion of 1 g ceftriaxone.
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | 150 mg SYN-004
Number analyzed (Participants) | 14
ug/mL
  Hour 0 | 0.00 (0.00)
  Hour 0.5 | 0.00 (0.00)
  Hour 1.5 | 9.80 (8.43)
  Hour 2.5 | 31.70 (22.57)
  Hour 3.5 | 42.80 (30.44)
  Hour 4.5 | 80.50 (56.28)
  Hour 5.5 | 0.80 (0.63)
  Hour 6.5 | 0.10 (0.10)
  Hour 7.5 | 0.00 (0.00)
  Hour 8.5 | 0.20 (0.14)

4. Primary Outcome: Ribaxamase Concentration in Intestinal Chyme Period 2
Description: Concentrations of ribaximase (SYN-004) in intestinal chyme
Time Frame: 0-8.5 hours
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | 150 mg SYN-004
Number analyzed (Participants) | 14
ng/mL
  Hour 0 | 0.00 (0.00)
  Hour 0.5 | 436 (435.6)
  Hour 1.5 | 281 (206.6)
  Hour 2.5 | 97745 (74180.)
  Hour 3.5 | 66936 (46358.5)
  Hour 4.5 | 63696 (26962.2)
  Hour 5.5 | 42316 (15114.4)
  Hour 6.5 | 38874 (21552.0)
  Hour 7.5 | 34756 (19642.6)
  Hour 8.5 | 35092 (20734.9)

ADVERSE EVENTS:
Groups:
- Treatment Period 1: In Treatment Period 1 (ceftriaxone + SYN-004), all 15 enrolled subjects received 1 g ceftriaxone and 14 received both 150 mg doses of SYN-004. One subject received only one 150 mg dose of SYN-004. In Treatment Period 1, one subject was discontinued from the study prior to receiving the second dose of SYN-004 due to a stoma site hemorrhage. The subject did not continue into the run-in phase or Treatment Period 2.
- Run-in Period: Treatment Periods 1 and 2 were separated by a 5- to 7-day run-in phase, during which subjects self-administered 40 mg of esomeprazole once daily in the morning.
- Treatment Period 2: In Treatment Period 2, subjects received 2 oral doses of 150mg SYN-004 and 1g ceftriaxone in the presence of esomeprazole. In Treatment Period 2 (ceftriaxone + SYN-004 + esomeprazole), 14 subjects were exposed to ceftriaxone, SYN-004, and esomeprazole. One subject did not receive study drug according to protocol.
Arm/Group | Treatment Period 1 | Run-in Period | Treatment Period 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/15 | 3/14 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period 1 (N=15) | Run-in Period (N=14) | Treatment Period 2 (N=14)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Stoma site hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators do not see trial results ahead of public disclosure unless it is under CDA. Investigators will not be allowed to publish or disclose any study results prior to sponsor communicating it to the public.